CLINICAL TRIAL: NCT06340451
Title: A Multicenter, Randomized, Double-Blind, Sham-Controlled Study Assessing the Efficacy and Safety of Iovera®° System in Subjects With Upper Extremity Spasticity
Brief Title: Study to Assess the Efficacy and Safety of Iovera®° System in Subjects With Upper Extremity Spasticity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IOV-301
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-10

CONDITIONS: Spasticity, Cerebral or Spinal Condition
Keywords: spasticity; cerebral; Spinal
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iovera° system treatment (Active Comparator)
  Interventions: Device: iovera° system
- sham iovera° system treatment (Sham Comparator)
  Interventions: Device: sham iovera° system treatment

INTERVENTIONS:
Device: iovera° system — subjects will receive ultrasound-guided iovera° system treatment
  Arms: iovera° system treatment
Device: sham iovera° system treatment — subjects will receive ultrasound-guided iovera° sham system treatment
  Arms: sham iovera° system treatment

SUMMARY:
This multicenter, randomized, double-blind, sham-controlled study is designed to evaluate the efficacy and safety of the iovera° system in subjects with upper extremity spasticity. A total of approximately 132 subjects will be enrolled; 88 subjects will receive treatment with the iovera° system and 44 subjects will receive sham treatment (sham iovera° system treatment).

DETAILED DESCRIPTION:
The screening and treatment may occur on the same day or be separated by as much as 30 days. All screening procedures must be completed, and criteria must be met before a subject is randomly assigned in the study. After random allocation to treatment, the subject will be scheduled for treatment (Day 1).

For all subjects, a Baseline (Day 1, pretreatment) Modified Ashworth Scale (MAS) score, Modified Tardieu Scale, and Goal Attainment Scale (GAS) score will be assessed and recorded before treatment on Day 1 (treatment day).

On Day 1 (treatment day), subjects will be reassessed for eligibility and randomly assigned in a blinded fashion (2:1) to receive either the iovera° system treatment or sham treatment. The study device will be used per the iovera° system User Guide on subjects who are prepared with local anesthetic (lidocaine 1%) only.

Local anesthetic will be injected subcutaneously into the treatment area. Ultrasound guidance will then be used to identify the specific target nerves to be studied. The targets of treatment are the medial and lateral pectoral nerves, and musculocutaneous nerve (motor branches to brachialis, and biceps brachii). A catheter will be used to guide the device needle. All subjects will have all target nerves treated. Nerve stimulation will also be employed as needed to assist in making an accurate determination regarding the location of the target nerves of interest. Up to two unblinded (1 primary and 1 backup) study staff (trained in the iovera° system treatment under ultrasound guidance) will be assigned per site to perform the study treatment procedures unless approved in advance in writing by the Sponsor on a case-by-case basis. The designated unblinded study staff must not participate in any other study-related assessments following treatment.

Each subject will be followed for 13 weeks post-treatment. The follow-up visits will be conducted at Week 3/Day 21 (±3), Week 7/Day 49 (±3), and Week 13/Day 91 (±5). Subjects will be assessed for efficacy and safety outcomes parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years and above.
2. A confirmed diagnosis of any cerebral or spinal condition, at least 6 months before Screening, resulting in spasticity of the muscles controlling the shoulder and elbow.
3. Not on oral medications for spasticity management or if on any oral medications, the oral medication taken chronically for spasticity management (eg, oral baclofen) must be maintained at a stable dose for at least 4 weeks before screening for the study.
4. Not on an intrathecal baclofen pump or if on an intrathecal baclofen pump for spasticity management, must be maintained at a stable dose for six months or more before screening for the study.
5. Must have a score on the Modified Ashworth Scale of 2 or more in the targeted area (shoulder and elbow) at Screening and at Baseline (Day-1 pretreatment).
6. A diagnostic nerve block using lidocaine (1% lidocaine, 2 to 3 mL per target nerve) showing a positive response (at least one point reduction from the screening Modified Ashworth Scale score for elbow extension and shoulder abduction) to the targeted nerves, should be performed within 30 days to at least 6 hours before study treatment. The diagnostic nerve block effect must be completely resolved before pretreatment evaluation and the study treatment.
7. Subject, in the investigator's opinion, will not be exposed to unacceptable risk by participation.
8. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. History of stroke, traumatic brain injury, and/or spinal cord injury in less than 6 months.
2. Diagnosis of cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, or Raynaud's disease.
3. History of neurotoxin injections within the past 3 months.
4. Previous injection with phenol or ethyl alcohol at any time in the target areas (shoulder or elbow).
5. Previous surgical intervention that altered the target neuroanatomy of the upper limb.
6. Current or planned enrollment in an investigational drug or device study for the management of spasticity for the duration of the study.
7. Medical instability that interferes with tolerability to spasticity treatment with the study device as per the investigator's discretion.
8. Any hospitalization within 4 weeks before Screening
9. Diagnosis of amyotrophic lateral sclerosis or any lower motor neuron conditions
10. Allergy or intolerance to amide local anesthetics.
11. Any skin condition in or around the target area that, in the opinion of the investigator, could adversely impact treatment.
12. Currently pregnant, nursing, or planning to become pregnant during the study.
13. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
14. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance.
15. Subject, in the opinion of the investigator, is not a suitable candidate for study participation (eg, history of multiple missed office visits, any related upper limb injury).
16. Subject is unable to adhere to the assessment schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Modified Ashworth Scale score for elbow measured (0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity) | at week 13

SECONDARY OUTCOMES:
Change from baseline in the Modified Ashworth Scale) score for shoulder (shoulder abduction) measured | at week 13
Change from baseline in the Modified Tardieu Scales for elbow (0 to 5, where lower score represents no resistance, and higher score represents joint immobility; Increase in angle from baseline [R1, and R2] represents improvement) | at week 13
Change from baseline in the Modified Tardieu Scales for shoulder (shoulder abduction) | at week 13
Change from baseline in Goal Attainment Scale score evaluated by the blinded, trained, licensed medical staff (-2 to +2, where lower score represents less expected outcomes, and higher scores represent greater expected outcomes) | at week 13

OTHER OUTCOMES:
Change from baseline in the Modified Ashworth Scale score for elbow measured immediately (within 3 hours) | at Day 1 post-treatment, Week 3, and Week 7
Change from baseline in the Modified Ashworth Scale score for shoulder (shoulder abduction) measured immediately (within 3 hours) | at Day 1 post-treatment, Week 3, and Week 7
Change from baseline in the Modified Ashworth Scale score for shoulder (forward flexion, external rotation) measured immediately (within 3 hours) | at Day 1 post-treatment, Week 3, and Week 7
Change from baseline in the Modified Ashworth Scale score over 13 weeks post-treatment measured by area under the curve (AUC) for elbow (elbow extension) | at week 13
Change from baseline in the Modified Ashworth Scale score over 13 weeks post-treatment measured by AUC for shoulder (shoulder abduction, shoulder forward flexion, external rotation) | at week 13
Change from baseline in the Modified Tardieu Scales for elbow measured immediately (within 3 hours) | at Day 1 post-treatment, Week 3, and Week 7.
Change from baseline in the Modified Tardieu Scales for shoulder (shoulder abduction) measured immediately (within 3 hours) | at Day 1 post-treatment, Week 3, Week 7, and Week 13
Change from baseline in the Modified Tardieu Scales for shoulder (forward flexion, external rotation) measured immediately (within 3 hours) | at Day 1 post-treatment, Week 3, Week 7, and Week 13
Change from baseline in Goal Attainment Scale score evaluated by the blinded, trained, licensed medical staff | at Week 3, and Week 7

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Source Healthcare - Santa Monica, Santa Monica, California
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Sarasota Memorial Hospital (SMH), Sarasota, Florida
  - Shepherd Center, Atlanta, Georgia
  - Kansas Institute of Research - Kansas City Bone & Joint Clinic, Overland Park, Kansas
  - University of Missouri Health Care - University Hospital, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper University Healthcare, Camden, New Jersey
  - Mount Sinai Health System - Faculty Practice Associates (FPA), New York, New York
  - Moss Rehab Physical Medicine Associates, Elkins Park, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) - Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Houston/TIRR, Houston, Texas
  - Virginia iSpine Physicians, PC, Richmond, Virginia
  - St. Luke's Rehabilitation Institute/Main Campus, Spokane, Washington
  - Center for Neurological Disorders - Gamma Therapeutic Center, Greenfield, Wisconsin
  - Froedtert and Medical College of Wisconsin - Milwaukee, Milwaukee, Wisconsin